CLINICAL TRIAL: NCT02324036
Title: The EMPATHy Toolkit: Helping Diabetes Patients Overcome Barriers to Medication Adherence
Acronym: EMPATHy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, John Thomas Billimek, Assistant Adjunct Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-1442
Record Dates: First submitted 2014-12-16; First posted 2014-12-24 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coached Care+EMPATHy; (Experimental): EMPATHy Toolkit: Patient coaching with computer assisted preference assessment
  Interventions: Device: EMPATHy Toolkit
- Routine Coached Care (Active Comparator): Patient coaching only
  Interventions: Behavioral: Coached Care

INTERVENTIONS:
Device: EMPATHy Toolkit — Software-based toolkit to help patients identify and prioritize barriers to medication adherence; community health worker provides participation training to patient
  Arms: Coached Care+EMPATHy;
Behavioral: Coached Care — Community health worker provides participation training to patient
  Arms: Routine Coached Care

SUMMARY:
The proposed study is a pilot study to gather data on the effectiveness and feasibility of a software tool (EMPATHy) to help patients communicate effectively with doctors about problems they face with their medication regimens. EMPATHy will be incorporated into an existing clinic-based intervention called Coached Care, in which community health workers (CHWs, non-professional community members) work as a "Coach" to patients to help them improve engagement and communication during the medical visit.

DETAILED DESCRIPTION:
Low income, Mexican American patients with diabetes exhibit high rates of medication nonadherence, which results in poor blood sugar control and serious complications, and often have difficulty communicating their concerns about the medication regimen to physicians. Interventions led by community health workers (CHWs), non-professional community members who are trained to work with patients to improve engagement and communication during the medical visit, have had mixed success in improving outcomes. Although CHWs possess excellent cultural competency and are very effective at establishing rapport with patients, they often lack a sophisticated understanding of all the potential challenges that can come with following a regimen. The primary objective of this project is to develop and pilot test a prototype software toolkit called "EMPATHy" that a CHW can administer to help patients identify and articulate the most important barriers to adherence that they face.

The EMPATHy toolkit will be piloted in an ongoing intervention (Coached Care) in which CHWs are trained to be "Coaches" to meet with patients before the medical visit, and help them prepare a list of important questions for the doctor. The Lead Researcher (Billimek) is a co-director of this intervention program at UCI's Ambulatory Clinics, including the Family Health Center in Santa Ana ,with a highly vulnerable population-low income Mexican American patients with diabetes and a history of nonadherence. A CHW will be trained to use two commercially available software programs configured by the PI to deliver the intervention materials. Patients participating in Coached Care (which is a clinic- based intervention, not a research protocol) will be recruited to (1) complete a Coached Care intervention session that has been modified to incorporate the EMPATHy Toolkit, (2) answer questions about barriers to medication adherence and the feasibility/usability of the software (3) allow the research team to abstract data on the medication regimen and diabetes outcomes (hemoglobin A1c, LDL cholesterol, etc) from the patient's medical record.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited from the University of California Irvine Federally Qualified Health Center family medicine clinic sites in Santa Ana and Anaheim with the following inclusion criteria:

  1. age 18 and older;
  2. have poorly controlled type 2 diabetes (as indicated by HbA1c>7.5%, LDL cholesterol >100 mg/dl or systolic blood pressure > 140),
  3. be of Hispanic ethnicity,
  4. speak English or Spanish.

These data are available to the research team in an automated report emailed to the lead researcher every week in his role as coordinator of the routine care Coaching program. This report includes a list of upcoming appointments for patients who meet these inclusion criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Development of a contextualized plan of care (assessed by analyzing an audio recording of the medical visit) | Baseline
  Development of a contextualized plan of care will be assessed by analyzing an audio recording of the medical visit, using a previously developed coding scheme (see Research Methodology). If the coder concludes that the plan of care discussed in the visit adequately addresses a contextual factor raised during the visit, it will be determined that a contextualized plan of care was developed.
Attainment of concrete behavioral goal (assessed in a two-week follow-up phone call to the patient) | 2 weeks post visit
  Attainment of concrete behavioral goal will be assessed in a two-week follow-up phone call to the patient, and will be defined as the patient reporting having completed the specific action that he or she specified with the Coach as a concrete goal during the intervention post-visit.

SECONDARY OUTCOMES:
Discussion of a contextual factor in the visit (assessed from audio recordings of the visit) | Baseline
  Discussion of a contextual factor in the visit will be assessed from audio recordings of the visit using a previously developed coding scheme. If the coder concludes that a relevant barrier to the patient taking his or her medication consistently was raised during the visit, it will be determined that a contextual factor was discussed.
Improvement in "red flag" outcome (assessed from the patient's medical record as the change in the measured value of the outcome measure identified as a high priority outcome) | 6 months post visit
  Improvement in "red flag" outcome will be assessed from the patient's medical record as the change in the measured value of the outcome measure identified as a high priority outcome ("red flag") from intervention visit date till the next regularly scheduled assessment. The red flag outcome measure is selected by the Coach and patient during the intervention visit, and can be either hemoglobin A1c, LDL cholesterol or blood pressure level.

CONTACTS AND LOCATIONS:
Overall Officials: John Billimek, PhD, Principal Investigator — Irvine
Locations (1):
- Health Policy Research Institute, Irvine, California, United States

REFERENCES:
- [Background] Billimek J, Guzman H, Angulo MA. Effectiveness and feasibility of a software tool to help patients communicate with doctors about problems they face with their medication regimen (EMPATHy): study protocol for a randomized controlled trial. Trials. 2015 Apr 10;16:145. doi: 10.1186/s13063-015-0672-7. PMID 25873349